CLINICAL TRIAL: NCT07017556
Title: An Exploratory Mixed-Methods Pilot Study on the Use of Educational Videos to Improve Knowledge and Satisfaction in Kidney Transplantation Patients
Brief Title: Views on Information Resources for Kidney Transplantation Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Responsible Party: Principal Investigator, Darren Manden, Principal Investigator, University of Auckland, New Zealand
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: KTPR2025
Record Dates: First submitted 2025-05-26; First posted 2025-06-12 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: End-Stage Renal Disease
Keywords: mixed-methods; pilot study; education; end-stage renal disease; kidney transplantation; feasibility study; repeated measures; video-based education; kidney disease
MeSH Terms: conditions — Kidney Failure, Chronic; Kidney Diseases

STUDY DESIGN:
Intervention Model Description: This study uses a single educational intervention across all participants. Participants are recruited from two subgroups:
  1. Pre-transplant patients - Recruited from the kidney transplant waitlist.
  2. Post-transplant patients - Recruited from post-transplant clinics.
  All participants receive the same educational resources (two short videos explaining the risks and benefits of kidney transplantation). The only difference between the subgroups is their transplant status, otherwise the intervention is the same for everyone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Video-Based Education (Pre / Post Transplant Patients) (Experimental): The study uses a single educational intervention for all participants. Participants are recruited from two subgroups: Pre-transplant patients, and post-transplant patients.
  All participants will watch the same educational videos (2 videos, each under five minutes) explaining important kidney transplant risks and benefits. These videos are designed to support the standard written and verbal information that patients receive.
  Information will be collected from participants at three time points:
  T1 (Day 1) - Immediately pre-video viewing. T2 (Day 1) - Immediately post-video viewing (the investigators will also conduct a short interview at this point).
  T3 (Day 7) - One week follow-up.
  Participants' knowledge and satisfaction will be assessed at each time point. Participants will also be interviewed to allow us to better understand their opinions. Analysis will examine differences by transplant status, but participants receive the same intervention.
  Interventions: Behavioral: Views on Information Resources for Kidney Transplantation Patients

INTERVENTIONS:
Behavioral: Views on Information Resources for Kidney Transplantation Patients — A pilot study to improve kidney transplant patient education. The study explores whether videos help patients to better understand and remember important information regarding the benefits and risks of receiving a kidney transplant.
  Currently, patients receive transplant information through written materials, and clinician discussions. However, not everyone has the same level of language literacy and medical understanding, which can lead to critical knowledge gaps, misunderstandings, and misinterpretations.
  Patients may also not know about lifelong medication needs, and complications which may follow transplantation, such as diabetes, making patient education and understanding essential.
  This study explores whether video materials helps patients feel more informed and satisfied with the clinical information they receive, and whether they can better retain this information. The investigators aim to support more informed patients, making transplant education clearer, and accessible.

SUMMARY:
The goal of this pilot study is to find out whether educational videos can help patients better understand, and remember, important information regarding the benefits and risks of having a kidney transplant.

The study aims to answer several questions, including:

1. Is the video-based educational intervention acceptable and feasible for kidney transplant patients?
2. Does the intervention improve patient knowledge and satisfaction immediately after viewing?
3. Does the intervention improve patient knowledge retention a week later?
4. What are patients views on the video format as an educational tool?

At the moment, patients learn about kidney transplantation through written documents, and discussions and conversations with their clinicians / doctors. However, the concern here is that not everyone has the same level of understanding when it comes to language literacy, medical jargon and information. This can result in gaps in knowledge, misunderstandings, and / or misinterpretations, including the need for lifelong medication and possible post-transplant complications.

Patients understanding of the benefits and risks of transplantation is extremely important, as there are aspects which patients may not be aware of, including the need for (and importance of) lifelong medication, and also potential disease complications which may follow transplantation. For example, following a kidney transplant, it is not uncommon for patients to develop diabetes.

Participants in the study will:

Watch two short videos (roughly five minutes each) that explain the benefits and risks of kidney transplantation.

Answer some questions before video viewing, immediately after video viewing, and one week after video viewing.

Complete a short interview to give deeper feedback on the videos.

This study will explore whether using video helps patients to feel more informed and also satisfied with the clinical information they receive, and whether they can better retain this information. The investigators aim to support more informed patients, making transplant education clearer, more accessible, and generally easier to understand.

DETAILED DESCRIPTION:
This will be a mixed-methods, repeated-measures, non-randomised pilot study. The design uses both quantitative and qualitative components to explore the feasibility and effectiveness of short (approximately five minutes each) educational videos for improving kidney transplant patient knowledge, knowledge retention, and information satisfaction.

A power analysis was conducted using G-Power to determine the participant sample size necessary for detecting a meaningful within-group effect of the intervention for both patient knowledge and information satisfaction. To detect a medium effect size (f = 0.21) with a power of 0.80 and an alpha level of .05, a total sample size of 60 participants (30 pre-transplant, and 30 post-transplant) is required.

Two subgroups (30 people each) - pre-transplant and post-transplant patients - will receive the same intervention with data collected through questionnaires (assessing knowledge, knowledge retention and satisfaction with the educational information) at three time points: Immediately pre-intervention (T1), immediately post-intervention (T2), and at a one-week follow-up (T3).

A semi-structured interview will take place immediately following the intervention (T2) exploring participants qualitative impressions of the videos and participant's assessment of the video's acceptability and the usefulness of the format.

The study will help to determine whether video-based education is a feasible and acceptable method for delivering kidney transplantation information, and whether it can improve participant understanding and satisfaction over traditional educational formats. The findings can then inform the design of a future larger-scale trial.

ELIGIBILITY:
Inclusion Criteria:

* Pre-transplant patients are on the kidney transplant wait list
* Post-transplant patients have received a transplant within the last 12 months.
* Participants are 18 years or over.
* Participants can read and understand English.
* Participants are located within the Auckland Metro region.

Exclusion Criteria:

* Any impairments preventing informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction with existing educational information | T1 - Day 1 (Immediately pre-video viewing).
  The Satisfaction with Existing Information questionnaire will be used to assess participants' satisfaction with the existing information received from their kidney transplant team. This will be used to help assess participants baseline satisfaction with standard kidney transplant education materials.
Patient understanding of kidney transplantation benefits and risks - Benefits | Patient understanding will be assessed at all three time points: T1 - Day 1 (Immediately pre-video viewing), T2 - Day 1 (Immediately post-video viewing), T3 - Day 7 (One week follow-up)
  One open-ended question will assess patient understanding of the benefits of kidney transplantation. This will be used to assess whether patient understanding of the benefits of transplantation changes from immediately pre-video viewing, to immediately post-viewing, and at one week follow-up.
Patient understanding of kidney transplantation benefits and risks - Risks | Patient understanding will be assessed at all three time points: T1 - Day 1 (Immediately pre-video viewing), T2 - Day 1 (Immediately post-video viewing), T3 - Day 7 (One week follow-up)
  One open-ended question will assess patient understanding of the risks of kidney transplantation. This will be used to assess whether patient understanding of the risks of transplantation changes from immediately pre-video viewing, to immediately post-viewing, and at one week follow-up.
Patient Satisfaction with video educational materials | T2 - Day 1 (Immediately post-video viewing), T3 - Day 7 (One week follow-up)
  The Satisfaction with Study Materials questionnaire will be used to assess participants' satisfaction with the video educational materials received from the research team. This will be used to assess participant satisfaction and to understand if the materials are coherent to participants, or if changes may be needed to make the materials more accessible, understandable, and effective.
Acceptability and usefulness of the study video resources (Qualitative) | T2 - Day 1 (Immediately post-video viewing).
  A semi-structured (15-20 minute) qualitative interview will take place at T2. This interview will explore patient thoughts of the materials beyond the questionnaires which they will receive. These interviews will explore participants' experience with the video material, including its perceived impact on benefits and risks understanding, and participant satisfaction with the Video-Based Educational materials - including acceptability, clarity and perceived usefulness. Interviews will explore suggestions for improving the intervention. Interview audio will be recorded and transcribed for thematic analysis.
Patient understanding of their disease | The BIPQ will be used at all three timepoints. T1 - Day 1 (Immediately pre-video viewing), T2 - Day 1 (Immediately post-video viewing), T3 - Day 7 (One week follow-up)
  The Brief Illness Perceptions Questionnaire (BIPQ) (Broadbent et al., 2006) will be used to assess participants' cognitive and emotional responses to their kidney transplantation; this will be used to help assess participants emotional response to both the risks and benefits of kidney transplantation.
Patient adherence to their medication | The AAI will be assessed at all three time points. T1 - Day 1 (Immediately pre-viewing), T2 - Day 1 (Immediately post-viewing), T3 - Day 7 (One week follow-up)
  The investigators will utilise questions from the Anticipated Adherence Index (AAI) (Wright, 2022) to identify if there is any change across timepoints for the participants views on the medication they are / will be taking, their intention to take their medication, and the importance of this medication to participants' long-term wellbeing.

CONTACTS AND LOCATIONS:
Overall Officials: Kate MacKrill, Dr, Principal Investigator — University of Auckland, New Zealand
Locations (1):
- Auckland City Hospital, Auckland, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
The investigators make available de-identified data available for Māori researchers upon reasonable request. Specifically: The investigators allow Māori organisations to access de-identified study data, for uses that may benefit Māori.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: By the time recruitment opens (estimated June 2025), and for no less than a year following publication of results.
Access Criteria: Māori researchers on reasonable request to the research team. People will receive a password protected Excel file containing the de-identified data.